CLINICAL TRIAL: NCT02573545
Title: Evaluation of a Support Software in the Planning and Real-time Monitoring of the Insertion of Needles in Interventional Magnetic Resonance Imaging (MRI): Liver Biopsy Case
Acronym: IFE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty recruiting patients
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 5261
Record Dates: First submitted 2015-10-01; First posted 2015-10-09 (Estimated); Last update posted 2019-12-04 (Actual); Status verified 2015-10

CONDITIONS: Liver Biopsy
Keywords: liver

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test group: with IFE (Experimental): Patients treated with IFE software
  Interventions: Device: Planning@IFE and Standard@IFE Software
- Test group: without IFE (Active Comparator): Patients treated with Numaris 4 software
  Interventions: Device: MR Syngo (Numaris/4) software

INTERVENTIONS:
Device: Planning@IFE and Standard@IFE Software
  Arms: Test group: with IFE
Device: MR Syngo (Numaris/4) software
  Arms: Test group: without IFE

SUMMARY:
To demonstrate that the use of Standard @IFE and Planning@IFE features of the IFE software, compared to the current method, when planning and inserting the needle under MRI monitoring in the context of liver biopsies enable:

* a facilitation of the planning stages of the procedure (route path, marking of the entry point and alignment of the MRI cutaways on the planned path), resulting in a reduction in the duration of the planning stages,
* a facilitation of the real-time modification of MRI cutaways during the procedure, resulting in a reduction of the duration of the procedure

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years old
* Affiliated to a social security scheme
* Informed consent
* Patient with an indication of liver biopsy eligible for a biopsy under interventional MRI

Exclusion Criteria:

* Patient with a contraindication for MRI exam
* Patient with a contraindication for performing a biopsy
* Pregnancy
* Exclusion period
* Patient unable to receive and understand information about the study
* Patients under guardianship
* Patients under judicial protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2013-01; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Total duration of the intervention (planning and implementation) | up to 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Nouvel Hôpital civil, Strasbourg, France